CLINICAL TRIAL: NCT04935554
Title: My Type 2 Diabetes: Person-centred Health Care
Acronym: MinT2D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Centre for Health Innovation (Unknown); The Dam Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 123998
Record Dates: First submitted 2020-10-22; First posted 2021-06-23 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Baseline testing with blood samples, blood pressure and 6 minute walking test. After answering a comprehensive screening tool questionnaire and a conversation with a resource person about "What is important to you", the study participant will chose one or several of the following interventions: physical activity, nutrition, motivation, health competence, psychosocial.
  Interventions: Other: Person centred care
- Control (No Intervention): Baseline testing with blood samples, blood pressure, 6 minute walking test and screening tool questionnaire.

INTERVENTIONS:
Other: Person centred care — physical activity, nutrition, motivation, health competence, psychosocial.
  Arms: Intervention

SUMMARY:
The Type 2 diabetes (T2D) project is a research and innovation project that will create a new comprehensive, participant-centered service model for interaction, increased physical activity, self-management, distance monitoring and lifestyle change for patients with type 2 diabetes. Central to the degree of innovation is a new model for interaction and use of technology for distance monitoring and coping.

DETAILED DESCRIPTION:
Type 2 diabetes is both physically and mentally stressful. At the same time, it requires a high individual effort, which can be demanding. Good mental health is necessary to be able to manage and control diabetes in a healthy and effective way. Therefore, we want to create an offer that takes care of the whole person, and physically as well as mentally.

Personal follow-up Based on surveys and conversations, the study participant and a contact person will prepare a 12-week plan that will be implemented with self-measurements and follow-up from the contact person. The plan will consist of the activities that best suit the participant's needs. It can be physical activity, diet course, health competence, motivation and psychosocial intervention that will be useful for the participant. After 12 weeks, the implementation will be evaluated.

Several new technological solutions are developed and will be used during the project period. A digital tool for mapping of the individuals needs will be an important part of the survey that is done during start-up. Activity clocks will be used for measuring steps, heart rate, and number of personalized activity index (PAI). An online portal for communication and interaction will make information easily accessible to users, simplify distance follow-up and communication flow.

The intervention will take place at two Healthy Life Centres. A Healthy Life Centre is an interdisciplinary primary health care service which offers effective, knowledge-based measures for people with, or in high risk of disease, who need support in health behaviour change and in coping health problems and chronic disease.

The Healthy Life Centre is part of the public health care service in the municipality. Healthy Life Centre programs have a patient centred approach and aim at strengthening the individual's control of his or her own health.

The intervention study starts in two municipalities in Møre og Romsdal, and the goal is to make the offer national.

ELIGIBILITY:
Inclusion Criteria:

• Type 2 diabetes

Exclusion Criteria:

* Unstable cardiovascular disease
* Severe chronic obstructive pulmonary disease (COPD)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Glycated haemoglobin (HbA1c) from baseline until week 12 | Baseline and week 12
  Glycated haemoglobin (HbA1c) is a measurement of the three-month average blood sugar level and HbA1c is an important outcome measure in diabetes clinical trials.

SECONDARY OUTCOMES:
Change in waist circumference from baseline until week 12 | Baseline and week 12
  Waist circumference is a simple method to assess abdominal adiposity that is easy to standardize and clinically apply. Waist circumference is strongly associated with all-cause and cardiovascular mortality
Change in physical fitness by the number of personalized activity index (PAI) from baseline until week 12 | Baseline and week 12
  Personalized activity index (PAI) was derived from an algorithm from one of the world's largest health studies (HUNT) and is a single, easy-to-understand personalized activity tracking metric that can help everyday people manage their health. Maintaining 100 PAI or more per week is strongly associated with adding on average 5 years to your life and reducing the risk of cardiovascular disease mortality by an average of 25%.
Health competence | Baseline and week 12
  The short version (HLS-Q12 ) of the European Health Literacy Survey Questionnaire (HLS-EU-Q47)
Change in mental health by questionnaire Symptom Checklist-90-R (SCL-90-R) until week 12 | Baseline and week 12
  The Symptom Checklist-90-R (SCL-90-R) is a relatively brief self-report psychometric instrument (questionnaire) published by the Clinical Assessment division of the Pearson Assessment & Information group. It is designed to evaluate a broad range of psychological problems and symptoms of psychopathology. SCL-90r is useful in measuring patient progress or treatment outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Ingul, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No